CLINICAL TRIAL: NCT05426005
Title: Cadonilimab (bispecific Anti-PD-1/CTLA-4 Antibody) for PD-1/PD-L1 Blockade-refractory, Microsatellite Instability-high (MSI-H) or Mismatch Repair-deficient (dMMR), Advanced Colorectal Cancer: a Single Group, Multicenter, Phase 2 Trial
Brief Title: Cadonilimab for PD-1/PD-L1 Blockade-refractory, MSI-H/dMMR, Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG-C03
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Stage IV; Mismatch Repair-deficient (dMMR); Microsatellite Instability-high (MSI-H)
Keywords: PD-1; CTLA-4; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Turcot syndrome; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadonilimab (Experimental): Cadonilimab alone
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab, 6 mg/kg every 2 weeks until disease progression, intolerable toxicity, or duration of treatment for 2 years

SUMMARY:
KEYNOTE-177 is currently the only randomized controlled phase III clinical trial evaluating the efficacy and safety of pembrolizumab versus standard chemotherapy combined with targeted first-line therapy for dMMR/MSI-H metastatic colorectal cancer. The study was conducted at 192 centers in 23 countries and enrolled a total of 307 subjects. The results of the study showed that the median PFS of pembrolizumab was 16.5 months, which was double the 8.2 months in the chemotherapy group (HR 0.60; 95% CI: 0.45-0.80; P = 0.0002). In addition, the ORR was 45.1% in the pembrolizumab group and 33.1% in the chemotherapy group, and a higher percentage of patients achieving a complete remission (CR) with pembrolizumab than in the chemotherapy group (13.1% vs. 3.9%). The U.S. FDA approved pembrolizumab in June 2020 for the first-line treatment of MSI-H/dMMR metastatic colorectal cancer.

The results of the KEYNOTE-177 study showed that 29% of patients with dMMR/MSI-H metastatic colorectal cancer experienced direct disease progression (PD) after first-line pembrolizumab monotherapy. This may suggest that some dMMR/MSI-H patients have primary resistance to anti-PD-1 monotherapy. In the first-line treatment cohort of the CheckMate 142 study using nivolumab combined with ipilimumab, the proportion of patients with direct PD was 13%, suggesting that the combination of PD-1 inhibitors and anti-CTLA-4 mAb may have help overcome this primary resistance. In addition, in the second-line and above cohort of the CheckMate142 study, 12% of patients receiving nivolumab in combination with ipilimumab experienced PD directly, compared with 26% of patients receiving nivolumab alone.

A study published on 《The Lancet Oncolog》 on the efficacy and safety of ipilimumab monotherapy and ipilimumab combined with anti-PD-1 monoclonal antibody in patients with anti-PD-1 monoclonal antibody-resistant melanoma Retrospective study. The study included 355 patients with unresectable metastatic stage III or IV melanoma who received ipilimumab monotherapy after failure of anti-PD-(L)1 monoclonal antibody (n=162), or Ipilimumab combined with anti-PD-1 therapy (n=193). The ORR was 31% in the combination arm, significantly higher than the 13% in the ipilimumab monotherapy arm. In addition, the median OS and PFS of the combination therapy group were 20.4 months and 3.0 months, respectively, which were also significantly higher than those of the single-agent group of 8.8 months and 2.6 months.

The aim of this study was to evaluate the objective response rate (ORR) of Cadonilimab, a bispecific anti-PD-1/CTLA-4 antibody, for PD-1/PD-L1 blockade-refractory, microsatellite instability-high (MSI-H) or mismatch repair-deficient (dMMR), advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Tumor tissues were identified as mismatch repair-deficient (dMMR) by immunohistochemistry (IHC) method or microsatellite instability-high (MSI-H) by polymerase chain reaction (PCR).
5. Subjects with stage IV colorectal cancer must have measurable or non measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.
6. Previous treatment with an anti-PD-1 or PD-L1 monoclonal antibody for advanced or metastatic colorectal cancer has failed. Treatment failure was defined as: disease progression or unacceptable toxicity during treatment or within 6 months after the last treatment.
7. Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.

Exclusion Criteria:

1. Previously received anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody.
2. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
3. Heart failure grade III/IV (NYHA-classification).
4. Unresolved toxicity higher than CTCAE v.5.0 Grade 1 attributed to any prior therapy/procedure.
5. Subjects with known allergy to the study drugs or to any of its excipients.
6. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
7. Breast- feeding or pregnant women.
8. Lack of effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
12-month Progression-free survival (PFS) rate | 2 years
  The PFS was defined as the time from enrollment until tumor progression or death from any cause, whichever occurred first. The 12-month PFS rate was defined as the proportion of patients without disease progression or death at the 12th month after initiation of the study. treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR).
Overall Survival (OS) | 5 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Toxicity assessed using the The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0. | 2 years
  The grade of toxicity will be assessed using the NCI-CTCAE, version 5.0. Grade refers to the severity of the AE. The CTCAE displays Grades 1 (lowest level) through 5 (highest level) with unique clinical descriptions of severity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China